CLINICAL TRIAL: NCT07109882
Title: Clinical Effectiveness of Chlorzoxazone Versus Orphenadrine Citrate in Alleviating Bruxism- Related Orofacial Pain: A Randomized Clinical Trial
Brief Title: Effectiveness of Chlorzoxazone Versus Orphenadrine Citrate in Alleviating Bruxism Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Noor R. Al-Hasani, Asst. Prof. Dr., University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1035425
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Orofacial Pain; Bruxism
MeSH Terms: conditions — Facial Pain; Bruxism | interventions — Chlorzoxazone; Orphenadrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorzoxazone Group (Active Comparator): Using Chlorzoxazone
  Interventions: Drug: Chlorzoxazone
- Orphenadrine Citrate group (Active Comparator)
  Interventions: Drug: Orphenadrine Citrate

INTERVENTIONS:
Drug: Chlorzoxazone — This group will receive Chlorzoxazone twice daily for two weeks
  Arms: Chlorzoxazone Group
Drug: Orphenadrine Citrate — This group will receive Orphenadrine Citrate twice daily for two weeks.
  Arms: Orphenadrine Citrate group

SUMMARY:
To evaluate the clinical effectiveness of chlorzoxazone in comparison to orphenadrine Citrate in relieving the orofacial pain in bruxers. Subjects and Methods: 60 patients above 15-years old complaining of orofacial and temporomandibular disorder/pain, with no history of chronic systemic illness, will be recruited. Patients will randomly be allocated into two groups (n=30): the first group will receive Relaxon (chlorzoxazone) twice daily for two weeks, while the second group will receive Norgesic (orphenadrine Citrate) twice daily for two weeks as well. Pain severity will be assessed by Visual Analogue Scale (VAS) at day 0, 7, and day 14. In addition, a temporomandibular joint (TMJ) evaluation form will be utilized to assess the TMJ parameters before and after initiation of the treatment protocol, i.e at 0 and 14 days. Non parametric statistical analysis will be conducted to explain the results using SPSS V29.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged above 15 years-old complaining of orofacial and temporomandibular disorder/pain.
* Patients with no history of chronic systemic illness.

Exclusion Criteria:

* Patients with orofacial injuries.
* Patients with head injuries.
* Patients Taking analgesics for the last 14 days.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Orofacial Pain Score in Bruxism Patients (n=30) as Measured by the Visual Analog Scale (VAS) in retaliation to adverse effect of each drug used. | From enrollment to the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Ameri LT, Issa SB, Abd Marzook A, Hameed EK, Jasem NH. Efficacy of Chlorzoxazone versus Orphenadrine in the management of pain associated with cervical spondylosis. Rawal Medical Journal. 2018;43:488-490.
- [Background] ElBohy D, Ateyya H, Elkot SM. Dentist & pharmacist communication awareness about skeletal muscle relaxants; survey in Egypt. Archives of Pharmaceutical Sciences Ain Shams University. 2023;7:240-253.
- [Background] Manfredini D, Lobbezoo F. Role of psychosocial factors in the etiology of bruxism. J Orofac Pain. 2009 Spring;23(2):153-66. PMID 19492540
- [Background] Bussadori SK, Motta LJ, Horliana ACRT, Santos EM, Martimbianco ALC. The Current Trend in Management of Bruxism and Chronic Pain: An Overview of Systematic Reviews. J Pain Res. 2020 Sep 30;13:2413-2421. doi: 10.2147/JPR.S268114. eCollection 2020. PMID 33061557
- [Background] Zielinski G, Pajak A, Wojcicki M. Global Prevalence of Sleep Bruxism and Awake Bruxism in Pediatric and Adult Populations: A Systematic Review and Meta-Analysis. J Clin Med. 2024 Jul 22;13(14):4259. doi: 10.3390/jcm13144259. PMID 39064299
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC7533232